CLINICAL TRIAL: NCT04115072
Title: Treatment of Female Genital Schistosomiasis (FGS) With Praziquantel: A Proof-of-Concept Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Regionshospital Nordjylland (Other Government)
Collaborators: Charite University, Berlin, Germany (Other); Leiden University Medical Center (Other); Nagasaki University (Other); Umeå University (Other); Merck Serono International SA (Industry); Ministry of Health, Madagascar (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHN_PCL_01
Record Dates: First submitted 2019-08-22; First posted 2019-10-03 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Praziquantel; Gynaecology; Female
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Single dose og PZQ (Active Comparator): Single dose of Praziquantel 40 mg/kg Standard treatment of schistosomiasis as recommended by WHO
  Interventions: Drug: Praziquantel 600Mg Oral Tablet x 1
- B - Five doses of PZQ (Experimental): Five doses of Praziquantel
  1 x 40 mg/kg Praziquantel after enrollment in the study plus two single doses (40 mg/kg) after 12 and 24 hours after the first treatment
  1 x 40 mg/kg Praziquantel five weeks following the 1st dose
  1 x 40 mg/kg Praziquantel ten weeks following the 1st dose
  Interventions: Drug: Praziquantel 600Mg Oral Tablet x 5

INTERVENTIONS:
Drug: Praziquantel 600Mg Oral Tablet x 5 — Five doses of Praziquantel 40 mg/kg
  Other Names: PZQ
  Arms: B - Five doses of PZQ
Drug: Praziquantel 600Mg Oral Tablet x 1 — Single dose of Praziquantel 40 mg/kg
  Other Names: PZQ
  Arms: A - Single dose og PZQ

SUMMARY:
Female genital schistosomiasis (FGS) is a frequent manifestation of the infection with Schistosoma haematobium or mansoni. FGS is probably the most neglected gynaecological condition in the tropics.

Inflammation of genital tissue persists as long as adult worms are present in the circulation, and new eggs are released. Hence, lesions can only heal if the inflammation is abated and a normal immune response is restored

A randomized controlled study will be carried out to compare the efficacy of the standard treatment with that of five repeated doses of praziquantel.

Outcome measure is the disappearance/regression of clinical pathology at the cervix, in the vagina/vulva.

DETAILED DESCRIPTION:
Female genital schistosomiasis (FGS) is a frequent manifestation of the infection with Schistosoma haematobium or mansoni. It occurs in women of all age groups, including young girls and is associated with important, frequently debilitating and stigmatizing morbidity. It may develop into a life-threatening condition. FGS is probably the most neglected gynaecological condition in the tropics.

Depending on where eggs are released the clinical pathology develops in vulva and vagina, cervix, uterus, Fallopian tubes and the ovaries. All genital organs may be affected simultaneously. Women with FGS report spontaneous, or post-coital bleeding, vaginal discharge, pain during sexual intercourse, pelvic pain, irregular menstruation and infertility. Vaginal discharge and itching, pain during sexual intercourse, spontaneous + post-coital bleeding, as well as menstruation abnormalities are attributed by the women to STIs. This results in shame, mental strain and distress, eventually causes stigmatization and social exclusion leading to an impaired life quality.

Clinical, histopathological, immunological and epidemiological evidence suggests that there is a cause-effect relationship between FGS and HIV infection. There are hints of a cause effect relationship between FGS and HPV. The association of FGS with HIV /HPV infection underlines the pivotal importance for an effective treatment of FGS.

Clinical pathology is the result of a complex inflammatory response to antigens released by adult worms and viable eggs. The inflammation of genital tissue persists as long as adult worms are present in the circulation, and new eggs are released and become trapped. Hence, lesions can only heal if the inflammation is abated and a normal immune response is restored. This means that all worms have to be eliminated and reinfection has to be prevented for some time to allow complete healing of genital organs.

Based on this rationale, five doses of praziquantel will be given over a period of 10 weeks to ensure that all existing worms will be eliminated. The first three doses aim to kill all adult worms. The fourth dose will kill schistosomula which will mature in the following weeks. The last dose will prevent women from re-infection.

A randomized controlled study will be carried out to compare the efficacy of the standard treatment with that of repeated doses of praziquantel. Since a placebo is not available, the study will not be blinded. Outcome measure is the disappearance/regression of clinical pathology at the cervix, in the vagina/vulva.

The result of this study has important implications for the sexual health of millions of women in sub-Saharan Africa.

The aim of the study is to compare standard treatment of schistosomiasis as recommended by WHO (a single dose of praziquantel 40 mg/kg)- with a treatment based on a new rationale: five doses of praziquantel 40 mg/kg

* 1 x 40 mg/kg after enrollment in the study (D1, H0) plus two single doses (40 mg/kg) after 12 and 24 hours after the first treatment
* 1 x 40 mg/kg five weeks following the 1st PZQ treatment
* 1 x 40 mg/kg ten weeks following the 1st PZQ treatment

ELIGIBILITY:
Inclusion Criteria:

* Women 15 to 35 years of age with a gynaecological/urinary/lower abdominal complaint
* The woman has signed the informed consent form (IFC); in the case of minors, the IFC has to be signed by parent or guardian.
* The woman does not plan to leave the area within 6 months and accept to come to the CSB regularly following the scheduled follow-up (at week 5,10 and 15).
* The woman with confirmed diagnosed of FGS (as described in section 6.3.1)
* The woman agrees to be examined clinically and gynaecologically including taking specimens from the genital tract (collection of vaginal lavage fluid, collection of cells with a cytobrush).
* The woman agrees to provide a urine and a stool sample.
* The woman agrees that a venous blood sample for laboratory assessments is taken.
* The woman accepts to stay at the hospital for 2 days follow-up after the first dose of PZQ.

Exclusion Criteria:

* Virgin (assessed by gynaecologist)
* Pregnancy (determined by pregnancy test)
* Tumor of vulva, vagina, uterus (diagnosed by gynaecologist)
* Treatment with praziquantel during the last 3 months
* Hysterectomy
* Known HIV positive prior to enrollment
* Any severe medical condition requiring hospitalization
* The woman is unable to comprehend the nature and objectives of the study
* The woman is judged by the investigators to be unlikely to participate regularly in the follow-up
* The woman is taking any drug that might affect the metabolism of PZQ and that is contraindicated the last two weeks before the enrollment. These drugs are as follows: rifampin; phenytoin, carbamazepine, phenobarbital; dexamethasone;
* The woman is taking a drug which decreases the activity of praziquantel metabolizing enzymes (P450 inhibitors) the last two weeks before the enrollment, for example cimetidine, ketoconazole, itraconazole, erythromycin.
* All contraindications to Praziquantel

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Pathognomonic sign(s) in the cervix | 15 weeks
  Changes is quantitatively measured by the comparison of the number of sectors of the cervix affected by a pathognomonic sign before treatment and at the end of the study.

SECONDARY OUTCOMES:
Gynaecological complaint score | 15 weeks
  Gynaecologial symptoms assessed by a questionnaire (Lower abdominal pain, Itching of vagina/vulva, Vaginal discharge with a strange odor, Pain/abnormal sensation during sexual intercourse, Bleeding after sexual intercourse, Abnormal sensation when touching vulva/vagina, Spontaneous bleeding (outside menstruation), Irregular menstruation, Infertility (primary or secondary) after two years without contraception, Pain during micturition, Blood in urine outside menstruation).
Vaginal Schistosome DNA | 15 weeks
  Concentration of schistosome DNA in vaginal fluid
Vaginal Pro-inflammatory Th2-dependent cytokines /chemokines | 15 weeks
  Concentration of selected pro-inflammatory Th2-dependent cytokines /chemokines in vaginal fluid
Vaginal ECP | 15 weeks
  Eosinophilic cationic protein (ECP) in vaginal lavage fluid
Cytobrush Schistosome DNA | 15 weeks
  Concentration of schistosome DNA in cytobrush material from vagina

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leutscher, PhD, Study Director — Centre for Clinical Research, North Denmark Regional Hospital, Denmark; Bodo S Randrianasolo, MD, Principal Investigator — K'OLO VANONA; Antananarivo, Madagascar
Locations (1):
- K'Olo Vanona, Ambanja, Diana Region, Madagascar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schuster A, Randrianasolo BS, Rabozakandraina OO, Ramarokoto CE, Bronnum D, Feldmeier H. Knowledge, experiences, and practices of women affected by female genital schistosomiasis in rural Madagascar: A qualitative study on disease perception, health impairment and social impact. PLoS Negl Trop Dis. 2022 Nov 7;16(11):e0010901. doi: 10.1371/journal.pntd.0010901. eCollection 2022 Nov. PMID 36342912
- [Derived] Arenholt LTS, Aaroe KK, Norderud K, Lumholdt M, Randrianasolo BS, Ramarokoto CE, Rabozakandraina O, Broennum D, Feldmeier H, Leutscher PDC. Cervical lesion proportion measure using a digital gridded imaging technique to assess cervical pathology in women with genital schistosomiasis. PLoS Negl Trop Dis. 2022 Jul 5;16(7):e0009995. doi: 10.1371/journal.pntd.0009995. eCollection 2022 Jul. PMID 35788749